CLINICAL TRIAL: NCT02445157
Title: Reliability of the 4 Metre Gait Speed in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Reliability of the 4 Metre Gait Speed in Idiopathic Pulmonary Fibrosis
Acronym: IPFREL
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14/LO/2248
Record Dates: First submitted 2015-05-01; First posted 2015-05-15 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Gait speed; Functional outcome measure
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IPF_Reliability: Patients diagnosed with IPF according to NICE guidelines.
  Interventions: Other: 4MGS

INTERVENTIONS:
Other: 4MGS — Measurement of usual gait speed over 4 metres (metres/second)
  Other Names: 4 metre gait speed test

SUMMARY:
This study is investigating the reliability of the 4 metre gait speed test (4MGS) in patients with a lung disease called Idiopathic Pulmonary Fibrosis (IPF).

DETAILED DESCRIPTION:
This observational study is investigating a simple test of walking speed, measured using the 4 metre gait speed test (4MGS), in patients with a lung disease called Idiopathic Pulmonary Fibrosis (IPF). Drug development for this disease is slow in part because there is a lack of reliable measurements that can assess effectiveness of treatment. Slow walking speed has been shown to relate to poor outcomes in older adults and people with another lung disease called Chronic Obstructive Pulmonary Disease (COPD. The investigators are interested to see whether usual walking speed is a reliable measure in patients with IPF as this will help inform us of its potential use as an outcome measure. To do this, participants who consent to taking part in the study will be timed walking at their usual walking speed over a distance of 4 metres (13.12 feet). Participants will be asked to do this twice with a rest in between if required. One week later, participants will be asked to repeat the walking tests again.

ELIGIBILITY:
Inclusion Criteria:

* IPF diagnosis according to NICE guidelines
* Provision of informed consent

Exclusion Criteria:

* Significant co-morbidities that would limit walking ability, exercise capacity or make exercise unsafe (e.g. unstable ischaemic heart disease, neuromuscular disease, severe hip/lower limb joint pain, peripheral vascular disease, lower limb amputation)
* Any patient whom the chief investigator feels it is unsafe to exercise (e.g. unstable cardiovascular disease)
* Any condition that precludes providing informed consent e.g. cognitive impairment or poor English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IPF according to NICE guidelines
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
4 metre gait speed | Change in gait speed measured at two timepoints one week apart
  Measure of usual walking speed

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, MD, PhD, Principal Investigator — Royal Brompton and Harefield NHS Foundtion Trust
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, Harefield, Middlesex, United Kingdom